CLINICAL TRIAL: NCT00860873
Title: Randomized Study of Two Dosage Forms (Oral Powder and Capsule) of "Chondroitin + Glucosamine Sulfate" Produced by the Laboratory EMS When Compared to the Product Condroflex (Oral Powder and Capsules) Produced by Laboratory Zodiac in the Treatment of Osteoarthrosis.
Brief Title: Effectiveness of Glucosamine + Chondroitin in Osteoarthrosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Azidus Brasil (Industry)
Responsible Party: Alexandre Frederico, LAL Clinica
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CGSEMS1108
Record Dates: First submitted 2008-11-26; First posted 2009-03-12 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Osteoarthrosis
MeSH Terms: conditions — Osteoarthritis | interventions — Glucosamine; Powders; Hardness

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Test 1 (Experimental): Oral Powder EMS
  Interventions: Dietary Supplement: EMS Chondroitin Sulfate + Glucosamine Sulfate (Oral powder)
- Test 2 (Experimental): Hard Capsules EMS
  Interventions: Dietary Supplement: EMS Chondroitin Sulfate 1200mg + Glucosamine Sulfate 1500mg (hard capsules)
- Comparator 1 (Active Comparator): Oral Powder Zodiac
  Interventions: Dietary Supplement: Zodiac: Chondroitin Sulfate 1200mg + Glucosamine Sulfate 1500mg (Oral powder)
- Comparator 2 (Active Comparator): Hard capsules - Zodiac
  Interventions: Dietary Supplement: Zodiac Chondroitin Sulfate 1200mg + Glucosamine Sulfate 1500mg (hard capsules)

INTERVENTIONS:
Dietary Supplement: EMS Chondroitin Sulfate + Glucosamine Sulfate (Oral powder) — Chondroitin Sulfate 1200mg Glucosamine Sulfate 1500mg
  Arms: Test 1
Dietary Supplement: EMS Chondroitin Sulfate 1200mg + Glucosamine Sulfate 1500mg (hard capsules) — Chondroitin Sulfate 1200mg Glucosamine Sulfate 1500mg
  Arms: Test 2
Dietary Supplement: Zodiac: Chondroitin Sulfate 1200mg + Glucosamine Sulfate 1500mg (Oral powder) — Chondroitin Sulfate 1200mg + Glucosamine Sulfate 1500mg
  Arms: Comparator 1
Dietary Supplement: Zodiac Chondroitin Sulfate 1200mg + Glucosamine Sulfate 1500mg (hard capsules) — Chondroitin Sulfate 1200mg + Glucosamine Sulfate 1500mg
  Arms: Comparator 2

SUMMARY:
This study objective is to check the non-inferiority of the 2 formulations produced by EMS when compared with the same substances and pharmaceuticals forms of the product Condroflex (Zodiac), by promoting the relief of osteoarthrosis symptoms such as pain, stiffness and functional capacity that will be periodically measured by using the "Visual Analog Scale" of pain (VAS) and the questionnaire of Lequesne.

ELIGIBILITY:
Inclusion Criteria:

* Patients who agree with all aspects of the study and sign the Informed Consent;
* Patients of both sexes;
* Age above 30 years;
* Clinical and radiological diagnosis of osteoarthritis;
* Osteoarthritis in grades 1-2;
* Patients who are conducting medical treatment and that, for trial of Investigator, is eligible for the study.

Exclusion Criteria:

* Patients with a history of trauma clinically significant;
* Patients who underwent surgery on joints affected;
* Coexistence of diseases that might impede the successful conclusion of the trial (rheumatism and others);
* Pregnant patients and / or breastfeeding;
* Patients with phenylketonuria;
* Patients with clinical diagnosis of severe renal failure;
* Patients with clinical diagnosis of severe liver disease;
* Patients with clinical diagnosis of clotting disorders;
* Patients who are being treated with anti-aggregating and / or anticoagulants;
* Patients with sensitive components of the formula;
* Patients with emotional disorders that interfere with the capture of data;
* Patients who do not agree with the purposes of the study and did not sign the Informed Consent.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2009-10; Primary Completion 2009-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Decrease in pain. | V0 (Screening); V1 (Inclusion); V2 (2 weeks); V3 (4 weeks); V4 (8 weeks); V5 (12 weeks); V6 (24 weeks).

CONTACTS AND LOCATIONS:
Locations (1):
- Lal Clinica Pesquisa E Desenvolvimento Ltda, Valinhos, São Paulo, Brazil